CLINICAL TRIAL: NCT01536405
Title: A Phase III Double-Blind, Randomized, Multicenter, Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of Measles, Mumps, Rubella, Varicella (MMRV) Vaccine Made With an Alternative Manufacturing Process (AMP)
Brief Title: Safety, Tolerability, and Immunogenicity of Measles, Mumps, Rubella, and Varicella (MMRV) Vaccine Made With an Alternative Manufacturing Process (AMP)(V221-027)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V221-027; P20930
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine; Adenosine Monophosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MMRV (AMP) (Experimental): Participants received two 0.5 mL subcutaneous injections of Mumps, Measles, Rubella, Varicella (MMRV) vaccine made with an alternative manufacturing process (AMP)
  Interventions: Biological: MMRV (AMP)
- MMRV (2006 process) (Active Comparator): Participants received two 0.5 mL subcutaneous injections of MMRV vaccine made with the 2006 manufacturing process
  Interventions: Biological: MMRV (2006 process)

INTERVENTIONS:
Biological: MMRV (AMP) — Measles, mumps, rubella, and VZV vaccine made with an alternative manufacturing process. Participants will receive two 0.5 mL subcutaneous injections.
  Arms: MMRV (AMP)
Biological: MMRV (2006 process) — Measles, mumps, rubella, and VZV vaccine made with the 2006 manufacturing process. Participants will receive two 0.5 mL subcutaneous injections.
  Other Names: ProQuad™
  Arms: MMRV (2006 process)

SUMMARY:
This study will compare the safety, tolerability, and immunogenicity of measles, mumps, rubella, and varicella (MMRV) vaccine made with an alternative manufacturing process with those of the 2006 process

ELIGIBILITY:
Inclusion Criteria:

* Negative clinical history for measles, mumps, rubella, varicella, and zoster

Exclusion Criteria:

* Received any measles, mumps, rubella, or varicella vaccine, either alone or in any combination at any time prior to the study, or is anticipated to receive any of these vaccines outside of study protocol, either alone or in any combination, during the study
* Received immune globulin, a blood transfusion or blood-derived products (does not include autologous blood/blood products) within 5 months (150 days) prior to any dose of the study vaccines or plans to receive these products while enrolled in this study
* Exposed to measles, mumps, rubella, varicella, or zoster within 4 weeks prior to the study vaccination
* Any congenital or acquired immune deficiency, neoplastic disease, or depressed immunity, including that resulting from steroid use or other immunosuppressive therapy
* Received 1) systemic immunomodulatory steroids [greater than the

equivalent of 2 mg/kg total daily dose of prednisone] within 3 months prior to

entering the study, or 2) any dose of systemic immunomodulatory steroids within

7 days prior to entering study, or 3) is expected to require systemic immunomodulatory steroids through the course of the study

* History of allergy or anaphylactoid reaction to gelatin, sorbitol, neomycin, egg proteins (eggs or egg products), chicken proteins, or any component of the study vaccines
* Received salicylates (eg, aspirin or aspirin-containing products) within 14 days prior to study vaccination
* Diagnosis of an active neurological disorder. Enrollment may be considered

when the disease process has been stabilized

* History of seizure disorder, including single febrile seizure
* Diagnosis of active untreated tuberculosis
* History of thrombocytopenia
* Born to a human immunodeficiency virus (HIV) infected mother

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1412 (Actual)
Dates: Start 2012-06-05 (Actual); Primary Completion 2013-07-02 (Actual); Study Completion 2014-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Marshall GS, Senders SD, Shepard J, Twiggs JD, Gardner J, Hille D, Hartzel J, Valenzuela R, Stek JE, Helmond FA. A double blind, randomized, active controlled study to assess the safety, tolerability and immunogenicity of measles, mumps rubella, and varicella vaccine (MMRV) manufactured using an alternative process. Hum Vaccin Immunother. 2016 Aug 2;12(8):2188-2196. doi: 10.1080/21645515.2016.1165374. Epub 2016 May 5. PMID 27149048
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V221-027&kw=V221-027&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was inadvertently randomized twice, for a total of 1413 randomizations. The Participant Flow reported below includes this participant only once.
Groups:
- MMRV (AMP): Participants were to received two 0.5 mL subcutaneous injections of Mumps, Measles, Rubella, Varicella (MMRV) vaccine made with an alternative manufacturing process (AMP)
- MMRV (2006 Process): Participants were to receive two 0.5 mL subcutaneous injections of MMRV made with the 2006 manufacturing process
Period: Randomization to Visit 1 (Vaccination 1)
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Started | 706 | 706
Completed | 698 | 702
Not Completed | 8 | 4
Not completed — Not vaccinated | 8 | 4
Period: Visit 1 (Vaccination 1) to Visit 2
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Started | 698 | 702
Received Vaccination 1 | 698 | 702
Completed | 666 | 662
Not Completed | 32 | 40
Not completed — Withdrawal by Subject | 12 | 18
Not completed — Lost to Follow-up | 20 | 22
Period: Visit 2 to Visit 3 (Vaccination 2)
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Started | 666 | 662
Completed | 635 | 634
Not Completed | 31 | 28
Not completed — Withdrawal by Subject | 17 | 13
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 9 | 10
Not completed — Protocol Violation | 2 | 2
Period: Visit 3 (Vaccination 2) to Visit 4
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Started | 635 | 634
Received Vaccination 2 | 634 | 632
Completed | 615 | 618
Not Completed | 20 | 16
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 16 | 14
Period: Visit 4 to Extended Study Follow-up
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Started | 615 | 618
Completed | 595 | 595
Not Completed | 20 | 23
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 20 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMRV (AMP) | MMRV (2006 Process) | Total
Number analyzed (Participants) | 706 | 706 | 1412
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.4 (2.2) | 13.6 (2.5) | 13.5 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 344 | 324 | 668
  Male | 362 | 382 | 744

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Varicella Zoster Virus (VZV) Antibody Levels >=5 gpELISA Units/mL
Description: Sera were tested for VZV Immunoglobulin (IgG) antibody levels by a glycoprotein enzyme-linked immunosorbent assay (gpELISA)
Time Frame: Six weeks after vaccination 1
Population: The per protocol population included participants who received >=1 dose of study vaccine, were seronegative at baseline and had postvaccination VZV serology results
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 586 | 589
Percentage of participants | 97.3 [95.6 to 98.4] | 93.0 [90.7 to 95.0]
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Non-Inferiority or Equivalence — The non-inferiority evaluation is based on the lower bound of the 2-sided 95% confidence interval (CI) on the risk difference excluding a decrease >= the prespecified criterion of 10 percentage points; p < 0.001, Miettinen and Nurminen; Risk Difference (RD) = 4.2, 95% CI 2-sided [1.8 to 6.8] — RD = MMRV (AMP) - MMRV (2006 process)
Statistical Analysis 2: Comparison: MMRV (AMP); Acceptability of the antibody response rate was based on a lower bound of the 95% CI being >76%; Test type: Superiority or Other; p < 0.001, One-sample binomial; Response rate = 97.3, 95% CI 2-sided [95.6 to 98.4]

2. Primary Outcome: Percentage of Participants With Measles Virus Antibody Levels >=255 mIU/mL
Description: Sera were tested for measles virus IgG antibody levels by an ELISA
Time Frame: Six weeks after vaccination 1
Population: The per protocol population included participants who received >=1 dose of study vaccine, were seronegative at baseline and had postvaccination measles virus serology results
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 629 | 621
Percentage of participants | 96.7 [94.9 to 97.9] | 98.9 [97.7 to 99.5]
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Non-Inferiority or Equivalence — The non-inferiority evaluation is based on the lower bound of the 2-sided 95% CI on the risk difference excluding a decrease >= the prespecified criterion of 5 percentage points; p = 0.003, Miettinen and Nurminen; Risk Difference (RD) = -2.2, 95% CI 2-sided [-4.0 to -0.6] — RD = MMRV (AMP) - MMRV (2006 process)
Statistical Analysis 2: Comparison: MMRV (AMP); Acceptability of the antibody response rate was based on a lower bound of the 95% CI being >90%; Test type: Superiority or Other; p < 0.001, One-sample binomial; Response rate = 96.7, 95% CI 2-sided [94.9 to 97.9]

3. Primary Outcome: Percentage of Participants With Mumps Virus Antibody Levels >=10 Units/mL
Description: Sera were tested for mumps virus IgG antibody levels by an enzyme-linked immunosorbent assay (ELISA)
Time Frame: Six weeks after vaccination 1
Population: The per protocol population included participants who received >=1 dose of study vaccine, were seronegative at baseline and had postvaccination mumps virus serology results
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 618 | 610
Percentage of participants | 98.2 [96.8 to 99.1] | 97.2 [95.6 to 98.4]
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; Risk Difference (RD) = 1.0, 95% CI 2-sided [-0.7 to 2.8] — RD = MMRV (AMP) - MMRV (2006 process)
Statistical Analysis 2: Comparison: MMRV (AMP); Acceptability of the antibody response rate was based on a lower bound of the 95% CI being >90%; Test type: Superiority or Other; p < 0.001, One-sample binomial; Response rate = 98.2, 95% CI 2-sided [96.8 to 99.1]

4. Primary Outcome: Percentage of Participants With Rubella Virus Antibody Levels >=10 International Units/mL (IU/mL)
Description: Sera were tested for rubella virus IgG antibody levels by an ELISA
Time Frame: Six weeks after vaccination 1
Population: The per protocol population included participants who received >=1 dose of study vaccine, were seronegative at baseline and had postvaccination rubella serology results
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 608 | 593
Percentage of participants | 98.8 [97.6 to 99.5] | 99.3 [98.3 to 99.8]
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; Risk Difference (RD) = -0.5, 95% CI 2-sided [-1.8 to 0.7] — RD = MMRV (AMP) - MMRV (2006 process)
Statistical Analysis 2: Comparison: MMRV (AMP); Acceptability of the antibody response rate was based on a lower bound of the 95% CI being >90%; Test type: Superiority or Other; p < 0.001, One-sample binomial; Response rate = 98.8, 95% CI 2-sided [97.6 to 99.5]

5. Primary Outcome: Geometric Mean Titer (GMT) of VZV Antibodies
Description: Sera were tested for VZV IgG antibody levels by gpELISA
Time Frame: Six weeks after vaccination 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 586 | 589
ELISA units/mL | 17.3 [16.4 to 18.3] | 14.4 [13.6 to 15.2]
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Non-Inferiority or Equivalence — The non-inferiority evaluation is based on the lower bound of the 2-sided 95% CI on the GMT ratio, excluding a decrease of >=1.5 fold; p < 0.001, t-test, 2 sided; Analysis was based on log-transformed titers; GMT ratio = 1.2, 95% CI 2-sided [1.1 to 1.3] — GMT ratio = MMRV (AMP) / MMRV (2006 process)

6. Primary Outcome: Geometric Mean Titer (GMT) of Measles Virus Antibodies
Description: Sera were tested for measles virus IgG antibody levels by ELISA
Time Frame: Six weeks after vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 629 | 621
mIU/mL | 3426.5 [3162.5 to 3712.4] | 3719.5 [3506.0 to 3946.0]
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 2 sided; Analysis was based on log-transformed titers; GMT ratio = 0.9, 95% CI 2-sided [0.8 to 1.0] — GMT ratio = MMRV (AMP) / MMRV (2006 process)

7. Primary Outcome: Geometric Mean Titer (GMT) of Mumps Virus Antibodies
Description: Sera were tested for mumps virus IgG antibody levels by ELISA
Time Frame: Six weeks after vaccination 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Mumps Ab units/mL
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 618 | 610
Mumps Ab units/mL | 112.1 [104.1 to 120.7] | 114.0 [105.8 to 122.8]
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 2 sided; Analysis was based on log-transformed titers; GMT ratio = 1.0, 95% CI 2-sided [0.9 to 1.1] — GMT ratio = MMRV (AMP) / MMRV (2006 process)

8. Primary Outcome: Geometric Mean Titer (GMT) of Rubella Virus Antibodies
Description: Sera were tested for rubella virus IgG antibody levels by ELISA
Time Frame: Six weeks after vaccination 1
Population: The per protocol population included participants who received >=1 dose of study vaccine, were seronegative at baseline and had postvaccination rubella virus serology results
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 608 | 593
IU/mL | 81.8 [76.8 to 87.2] | 80.7 [76.4 to 85.2]
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 2 sided; Analysis was based on log-transformed titers; GMT ratio = 1.0, 95% CI 2-sided [0.9 to 1.1] — GMT ratio = MMRV (AMP) / MMRV (2006 process)

9. Primary Outcome: Percentage of Participants With Fever (>=102.2°F [39.0°C] or Oral Equivalent)
Time Frame: Up to 5 days after vaccination 1
Population: The population analyzed included participants who received >=1 study vaccination and had follow-up safety data
Measure: Number; unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 645 | 648
Percentage of participants | 0.9 | 0.8
Statistical Analysis 1: Comparison: MMRV (AMP) vs MMRV (2006 Process); Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Risk Difference (RD) = 0.2, 95% CI 2-sided [-1.0 to 1.3] — RD = MMRV (AMP) - MMRV (2006 process)

10. Secondary Outcome: Percentage of Participants With Fever (>=102.2°F [39.0°C] or Oral Equivalent)
Time Frame: Up to 42 days after each vaccination
Population: The population analyzed included participants who received >=1 study vaccination and had follow-up safety data
Measure: Number; unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 650 | 649
Percentage of participants
  Vaccination 1; n=650, n=649 | 10.0 | 10.6
  Vaccination 2; n=592, n=597 | 5.7 | 8.4

11. Secondary Outcome: Percentage of Participants With Zoster-like Rash
Time Frame: Up to 42 days after each vaccination
Population: The population analyzed included participants who received >=1 study vaccination and had follow-up safety data
Measure: Number; unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 682 | 682
Percentage of participants
  Vaccination 1; n=682, n=682 | 0.0 | 0.0
  Vaccination 2; n=634, n=632 | 0.0 | 0.0

12. Secondary Outcome: Percentage of Participants With Mumps-like Symptoms
Time Frame: Up to 42 days after each vaccination
Population: The population analyzed included participants who received >=1 study vaccination and had follow-up safety data
Measure: Number; unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 682 | 682
Percentage of participants
  Vaccination 1; n=682, n=682 | 0.0 | 0.0
  Vaccination 2; n=634, n=632 | 0.0 | 0.0

13. Secondary Outcome: Percentage of Participants With Measles-like Rash
Time Frame: Up to 42 days after each vaccination
Population: The population analyzed included participants who received >=1 study vaccination and had follow-up safety data
Measure: Number; unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 682 | 682
Percentage of participants
  Vaccination 1; n=682, n=682 | 0.1 | 0.3
  Vaccination 2; n=634, n=632 | 0.2 | 0.0

14. Secondary Outcome: Percentage of Participants With Rubella-like Rash
Time Frame: Up to 42 days after each vaccination
Population: The population analyzed included participants who received >=1 study vaccination and had follow-up safety data
Measure: Number; unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 682 | 682
Percentage of participants
  Vaccination 1; n=682, n=682 | 0.0 | 0.0
  Vaccination 2; n=634, n=632 | 0.0 | 0.0

15. Secondary Outcome: Percentage of Participants With Varicella-like Rash
Time Frame: Up to 42 days after each vaccination
Population: The population analyzed included participants who received >=1 study vaccination and had follow-up safety data
Measure: Number; unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 682 | 682
Percentage of participants
  Vaccination 1; n=682, n=682 | 0.6 | 0.0
  Vaccination 2; n=634, n=632 | 0.0 | 0.0

16. Secondary Outcome: Percentage of Participants With an Injection-site Adverse Event
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Injection-site AEs reported were solicited with a Vaccine Report Card.
Time Frame: Up to 5 days after each vaccination
Population: The population analyzed included participants who received >=1 study vaccination and had follow-up safety data
Measure: Number; unit: Percentage of participants
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Number analyzed (Participants) | 682 | 682
Percentage of participants
  Vaccination 1; n=682, n=682 | 36.4 | 29.8
  Vaccination 2; n=634, n=632 | 35.5 | 29.6

ADVERSE EVENTS:
Time Frame: Up to 6 months (180 days) after vaccination 2
Description: The All Subjects as Treated population included randomized participants who received >=1 dose of study vaccine and had safety follow-up results
Arm/Group | MMRV (AMP) | MMRV (2006 Process)
Serious Adverse Events (participants affected / at risk) | 21/682 | 18/683
Other Adverse Events (participants affected / at risk) | 574/682 | 572/683
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMRV (AMP) (N=682) | MMRV (2006 Process) (N=683)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis staphylcoccal (Infections and infestations) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 2 (2)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0)
Exposure via direct contact (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure via ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 4 (5) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMRV (AMP) (N=682) | MMRV (2006 Process) (N=683)
Conjunctivitis (Eye disorders) | 48 (52) | 46 (47)
Diarrhoea (Gastrointestinal disorders) | 77 (98) | 91 (107)
Vomiting (Gastrointestinal disorders) | 60 (77) | 61 (72)
Injection site erythema (General disorders) | 254 (344) | 199 (258)
Injection site pain (General disorders) | 208 (267) | 187 (243)
Injection site swelling (General disorders) | 156 (190) | 123 (146)
Pyrexia (General disorders) | 225 (349) | 235 (360)
Gastroenteritis (Infections and infestations) | 29 (32) | 41 (43)
Nasopharyngitis (Infections and infestations) | 55 (65) | 66 (76)
Otitis media (Infections and infestations) | 128 (177) | 128 (179)
Otitis media acute (Infections and infestations) | 56 (72) | 44 (57)
Pharyngitis (Infections and infestations) | 40 (47) | 35 (43)
Upper respiratory tract infection (Infections and infestations) | 159 (210) | 163 (212)
Viral infection (Infections and infestations) | 44 (52) | 57 (64)
Cough (Respiratory, thoracic and mediastinal disorders) | 87 (113) | 101 (118)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 58 (78) | 53 (64)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 62 (76) | 77 (106)
Rash (Skin and subcutaneous tissue disorders) | 48 (50) | 47 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.